CLINICAL TRIAL: NCT04723654
Title: Evaluating Wearable Smart Sensors for Continuous Measurement of Vital Signs in ICU
Brief Title: Evaluating Wearable Smart Sensors for Continuous Measurement of Vital Signs in ICU Patients
Status: Recruiting | Type: Observational
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Susan Slattery, Attending Physician, Ann & Robert H Lurie Children's Hospital of Chicago
Other Study IDs: 2018-1668
Record Dates: First submitted 2021-01-13; First posted 2021-01-26 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Prematurity
Keywords: Blood Pressure; Vital Signs; Wireless Monitoring
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ICU Population: Patients admitted to one of 3 ICUs at Lurie Childrens
  Interventions: Device: Wireless Wearable Vital Sign Monitor
- Non-ICU Population: Healthy volunteers who are under 18 years of age, whose parents consent to their participation, and who are willing to visit CAMP for a one time study visit can participate in this study.
  Interventions: Device: Wireless Wearable Vital Sign Monitor

INTERVENTIONS:
Device: Wireless Wearable Vital Sign Monitor — Placement of wireless wearable vital sign monitors on patients limbs for up to 48 hours

SUMMARY:
The purpose of this study is to develop biocompatible wireless electronic devices that will allow continuous, non-invasive hemodynamic and physiology measurements in the ICU.

DETAILED DESCRIPTION:
Screening: All ICU patients will be screened by the study team based on inclusion and exclusion criteria through review of electronic medical records. For screening at Prentice Women's Hospital, screening criteria will be automatically applied through the use of the electronic data warehouse, and information from infants meeting this screening criteria will be transferred to the study team through electronic data warehouse. A screening and enrollment log will be kept to track ICU patients/parents who have been approached and agreed or declined to participate in the study. The screening and enrollment log will be kept on the Northwestern University housed REDCap server. Only the study team will have access to this log. All non-ICU participants will be screened through question and answer with a parent or guardian.

Device application: Standard devices will be used continuously in all subjects and this data compared to that collected using novel wearable sensors suggested in this study. In the ICU population, after patients are consented in the ICU, multiple wearable sensors (up to 5) will be placed on the patient for the duration of the study. Multiple devices are required to estimate BP. One or more devices will be placed on the chest or back, and one or more additional devices will be placed peripherally (e.g. leg, foot, arm, hand, head, or ear). Placing multiple devices will allow determination of which location provides the best signals in specific ICU populations. These devices will be placed using a medical grade skin adhesive similar to the ones used in the ICUs, which will minimize the risk of skin irritation or allergic reaction. Alternatively, the investigators are currently testing a "soft wrap-around device" (similar to that currently used for blood pressure monitoring in the premature babies) with a sensor. The soft wrap-around device is composed of hypoallergenic cotton. Overlying this cotton, and not touching the subject's skin, may include Coban wraps, paper tape, or a Velcro adhesion mechanism. Given the very small size of premature infants in the NICU, the investigators may incorporate this new technology as needed in the NICU. Each device is encapsulated in medical grade materials and applied using medical grade adhesive. The adhesives will be changed between uses. The device itself will be re-used. It will be cleaned with Super Sani-Cloth between each use. In the ICU population, devices will be left in place for up to 48 hours, but will be checked by study staff to ensure skin integrity and signal quality at least once every 24 hours. In the non-ICU population, standard of care devices will be attached to participants according to ICU standard of care procedures. The wearable sensors will be placed in the same manner as outlined above but will be left in place for only up to 3 hours during an outpatient study visit to the Center for autonomic Medicine in Pediatrics (CAMP).

The investigators have recently upgraded a new firmware version activating the ability for the sensor to continuously measure bioimpedance for respiratory rate. This function does not require any modification to the physical device itself or the adhesive. However, the bioimpedance functionality does require delivery of low amplitude sinusoidal current through the electrodes of the chest unit. The frequency of the current is 4 kHz - a frequency range used typically for human bioimpedance measurements by FDA cleared systems. The maximum current delivered is 8 μA. These parameters are below commonly used body fat percentage impedance analyzers that are widely commercially available. Furthermore, bioimpedance is standardly used in NICUs / PICUs leveraging the ECG electrodes that are then displayed on standard of care monitors. Commercially bioimpedance devices that are FDA approved inject currents that are 10x greater than our system (e.g. the CoVa Monitoring System 2 for continuous wearable sensing of thoracic impedance). Finally, the parameters in our sensor follow IEC 60601-1-2 guidelines for electromagnetic safety.

Video monitoring: In some participants, video monitoring of participant position and movement will be utilized during the study. This is an optional, additional part of the study in which families can choose to participate or not participate. If a family chooses to participate, a video camera will be utilized to capture participant movement and position for the duration of the study in the ICU or at CAMP.

Cuff-based blood pressure: While the wearable sensors are attached to participants in both the ICU and non-ICU populations, the participants will also be monitored with the normal standard of care monitoring montage. In addition, during one 3- or 4-hour period while the wearable sensors are attached to the patient, a member of the study team may take the participant's BP using the ICU standard cuff-based method every 15 minutes. Cuff-based measures typically happen every 15-60 minutes for standard clinical care, depending on the stability of the patient and physician discretion. In the ICU cohort, if a standard clinical cuff-based BP measure is taken during the 15-minute time epoch, the clinical measurements will be used rather than obtaining a separate research measurement. Outside of this 3- or 4-hour window and for the remainder of the study duration in the ICU population, cuff-based BP measures will be made only as frequently as needed for standard clinical care.

Skin temperature: While the wearable sensors are attached to the participant, skin temperatures will be taken using a standard infrared thermometer. These measurements will be made at the same interval as the above cuff-based BP, over the same 3- or 4-hour period by a member of the study team. Outside of this 3- or 4-hour window, no skin temperature measures will be made for research purposes.

Device data: Wearable sensors can stream data continuously using near field communication (NFC) or Bluetooth technology. An encrypted laptop, iPad, or similar device will be left in the patient or CAMP study room and used to capture the continuous data stream from the wearable sensor. Additionally, wearable sensors can include onboard memory, and physiologic streams may be recorded to this onboard memory until transfer to an encrypted laptop for analysis.

Standard of care data: In all participants where data from standard of care monitoring is captured and stored using the BedMasterEx system (all PICU and CCU beds, some NICU beds), these data will be used for comparison to data captured using EWP. In any participants where data are not captured and stored using the BedMasterEx system, video recordings will be made of the Phillips monitors using an encrypted mobile device. Within 48 hours, videos will be downloaded and transferred to a HIPAA secure server. In NICU patient without BedMasterEx data, the Somnostar system may be used to capture data for up to 4 hours of the study. All study data will be stored on an encrypted laptop and/or secure networkfor analysis.

Skin integrity: Before and after wearable sensors are placed on the participant, the participant's skin integrity will be monitored using the ICU standard protocol, either the Braden Q scale (≥6 months of age) and/or Neonatal Skin Risk Assessment Scale (NSRAS; <6 months of age). Additionally, a member of the study team will use a validated skin integrity scale to score participants' skin condition at sensor placement site before sensor placement and immediately after sensor removal. At both of these time points, photographs will be taken of the participants' skin at the site of sensor placement to document any skin changes that occur during the period of wearable sensor wear. No faces will be photographed. Additional skin scores and photographs may be performed/taken between 30 minutes and 24 hours after sensor removal, as deemed necessary by the study and/or clinical team. The study team will consult the ICU bedside care team or CAMP clinical team within 1 hour for any concerning changes in skin integrity.

Questionnaires: After the study period ends, the parents will be approached to complete the questionnaires. These questionnaires will take less than 10 minutes to complete and are meant to assess opinions on use of these devices in the ICUs. These questionnaires will be completed using REDCap or a printed version of the REDCap questionnaire. All questionnaire data will be stored on the secure REDCap server housed by Northwestern University.

ELIGIBILITY:
Inclusion Criteria-ICU Population:

* Admitted to one of the four ICUs at Lurie Children's or Prentice Women's Hospital
* Under 18 years of age

Inclusion Criteria-Non-ICU Population

* Under 18 years of age
* Willing to visit the Center for Autonomic Medicine in Pediatrics (CAMP) for a one time study visit

Exclusion Criteria-ICU Population:

* A skin abnormality that would potentially increase the risk of device
* 18 years of age or older
* Determined by an attending physician or bedside care team to be too unstable (patient) or experiencing too much stress (family)

Exclusion Criteria-Non-ICU Population:

* A skin abnormality that would potentially increase risk of device use
* 18 years of age or older

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients admitted to one of 3 ICUs at Lurie Children's, or healthy volunteers visiting CAMP at Lurie Children's
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-03-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Continuous non-invasive BP monitoring | up to 48 hours
  Recorded measurements of BP as compared to the ICU standard of care monitoring, including both arterial line measurements and cuff-based measurements of the arm (mm Hg).

SECONDARY OUTCOMES:
Accuracy of Other Physiologic Signals | up to 48 hours
  correlation of vital signs to current technology used on the units: heart rate (beats/min); respiratory rate (breaths/min); temperature (degrees Celsius); oxygen saturation (SpO2, %)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Northwestern Medicine Prentice Women's Hospital, Chicago, Illinois

REFERENCES:
- [Background] Chung HU, Rwei AY, Hourlier-Fargette A, Xu S, Lee K, Dunne EC, Xie Z, Liu C, Carlini A, Kim DH, Ryu D, Kulikova E, Cao J, Odland IC, Fields KB, Hopkins B, Banks A, Ogle C, Grande D, Park JB, Kim J, Irie M, Jang H, Lee J, Park Y, Kim J, Jo HH, Hahm H, Avila R, Xu Y, Namkoong M, Kwak JW, Suen E, Paulus MA, Kim RJ, Parsons BV, Human KA, Kim SS, Patel M, Reuther W, Kim HS, Lee SH, Leedle JD, Yun Y, Rigali S, Son T, Jung I, Arafa H, Soundararajan VR, Ollech A, Shukla A, Bradley A, Schau M, Rand CM, Marsillio LE, Harris ZL, Huang Y, Hamvas A, Paller AS, Weese-Mayer DE, Lee JY, Rogers JA. Skin-interfaced biosensors for advanced wireless physiological monitoring in neonatal and pediatric intensive-care units. Nat Med. 2020 Mar;26(3):418-429. doi: 10.1038/s41591-020-0792-9. Epub 2020 Mar 11. PMID 32161411
- [Background] Chung HU, Kim BH, Lee JY, Lee J, Xie Z, Ibler EM, Lee K, Banks A, Jeong JY, Kim J, Ogle C, Grande D, Yu Y, Jang H, Assem P, Ryu D, Kwak JW, Namkoong M, Park JB, Lee Y, Kim DH, Ryu A, Jeong J, You K, Ji B, Liu Z, Huo Q, Feng X, Deng Y, Xu Y, Jang KI, Kim J, Zhang Y, Ghaffari R, Rand CM, Schau M, Hamvas A, Weese-Mayer DE, Huang Y, Lee SM, Lee CH, Shanbhag NR, Paller AS, Xu S, Rogers JA. Binodal, wireless epidermal electronic systems with in-sensor analytics for neonatal intensive care. Science. 2019 Mar 1;363(6430):eaau0780. doi: 10.1126/science.aau0780. PMID 30819934

DOCUMENTS (1):
  • Study Protocol (2024-10-03): https://cdn.clinicaltrials.gov/large-docs/54/NCT04723654/Prot_001.pdf